CLINICAL TRIAL: NCT06160258
Title: Impact of Convenience on Consumption of Intact Novel Whole Grains: A Comparison Between Ready-to-Eat and Dried Conditions
Brief Title: Impact of Convenience on Whole Grain Consumption
Acronym: WG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lisa Grentz, Associate, Washington State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20358
Record Dates: First submitted 2023-11-28; First posted 2023-12-07 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Health Behavior; Diet, Healthy; Diet Habit
Keywords: whole grains; convenience; ready-to-eat
MeSH Terms: conditions — Health Behavior; Feeding Behavior | interventions — Fast Foods; Desiccation

STUDY DESIGN:
Intervention Model Description: The study employs a two-arm, randomized parallel design. Individuals, ages 19+, will be randomly assigned to one of two 4-week intervention conditions in which they receive either precooked intact novel whole grains ("RTE" condition) or dried, bulk novel whole grains ("DRIED" condition) to consume at home.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ready-to-Eat condition (Experimental): Participants will be provided precooked and individually packaged whole grains in the ready-to-eat condition for reheating and consumption at home.
  Interventions: Behavioral: Ready to Eat (RTE)
- Dried condition (Experimental): Participants will be provided with whole grains of barley, buckwheat, and quinoa in the dried, bulk condition for home cooking and consumption.
  Interventions: Behavioral: Dried

INTERVENTIONS:
Behavioral: Ready to Eat (RTE) — Participants will be provided precooked and individually packaged whole grains in the ready-to-eat (RTE) condition for reheating and consumption at home.
  Arms: Ready-to-Eat condition
Behavioral: Dried — Participants will be provided with dried whole grains for home preparation and consumption
  Arms: Dried condition

SUMMARY:
Intact whole grains (such as quinoa, buckwheat, and barley) contain all 3 parts of the kernel (bran, germ, and endosperm) compared to processed grains where the bran and germ layers have been removed. Intact whole grains have a higher nutritional value but are under consumed in the diet of most adults. In this proposed pilot study, 42 participants will be recruited to study the impact of convenience on intake of intact whole grains by comparing consumption of intact whole grains that are offered in a convenient pre-cooked ready-to-eat form compared to traditional bulk dried form that requires a more prolonged preparation and cooking time. The ready-to-eat meals will be processed using WSU microwave technologies to ensure food safety. All intact whole grains (ready-to-eat or dried) will be provided to participants, who will prepare and consume the grains at home over a period of 4 weeks. Type and volume of whole grain consumed will be monitored daily via REDCap survey, which will allow the investigators to see if adults are more likely to meet daily recommended intakes of whole grain servings when offered in a convenient form.

DETAILED DESCRIPTION:
The investigators will evaluate the effects of convenience on intake of intact whole grains. Forty-two participants (19 years or older) will be randomized to receive intact whole grains of barley, buckwheat, and quinoa in either a convenient ready-to-eat (RTE) form or a bulk (DRIED) form. Enrollment in the study will continue until 42 participants have completed the study. Recruitment will include posters, word-of-mouth, and online newsletters. Interested individuals will complete an online survey to determine initial eligibility. Eligible participants will be contacted by study staff and invited to an in-person orientation session. At the in-person visit, participant eligibility will be verified. Eligible participants will review and sign the informed consent form. Using standard clinical protocols, trained research staff will collect baseline measurements of height and weight, randomize participants to either the RTE or DRIED condition, provide education on whole grains and how to prepare the study grains, and provide participants with a link to complete a questionnaire about eating habits. Lastly, participants will be sent home with the 7 days' worth of study grains. This visit will take up to 90 minutes to complete.

The intervention is a total of four weeks, during which participants will incorporate intact whole grains into their usual diet. Four weeks should be a sufficient to observe dietary changes. Daily during the study, participants will be prompted to complete a brief online survey to report the type and amount of study grains consumed over the course of the day.

Once per week during the intervention, participants will visit the WSU Food Lab, located in the Health Sciences Building on the WSU - Spokane Campus, for a 10-15-minute visit. During each visit, the investigators will provide one weeks' worth of study grains and review adherence to study protocols. At the end of the fourth week, participants will return to the laboratory for a final exit visit where study staff will measure participant weight and administer an exit survey and food frequency questionnaire. Statistical power calculations indicate that forty-two participants included in this pilot study is sufficient for detecting an effect of whole grain intake between the two study conditions.

ELIGIBILITY:
Inclusion Criteria:

* Able to communicate in written and spoken English
* Not following a restricted diet
* Involved in home food preparation
* Daily access to working internet
* Daily access to working microwave, stove, refrigerator, and freezer

Exclusion Criteria:

* Dietary restrictions, including allergy/intolerances
* Latex allergy
* Following a diet to increase or decrease body weight
* Taking medications that promote weight loss
* Use of nicotine, marijuana, or illicit drugs
* Pregnancy, planned pregnancy, or breastfeeding
* Inability to comprehend the nature of the study instructions
* No access to internet
* Planning to leave the Spokane area during the study
* Not fluent in the English language

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Determine the effect of convenience on intake of intact cooked whole grains over a 4-week period | 4-week period
  Participants in the ready-to-eat condition and dried condition will self report type of cooked whole grain and quantity of cooked whole grains consumed daily in REDCap. The investigators will compare total intake of whole grains between the ready-to-eat and dried conditions as reported on daily REDCap checklists.

SECONDARY OUTCOMES:
Determine the effect of a dietary intervention on intake of whole grains over a 4-week period | 4-week period
  Compare baseline whole grain ounce equivalents to endpoint ounce equivalents using DHQIII.

CONTACTS AND LOCATIONS:
Overall Officials: Martine Perrigue, PhD, RD, Principal Investigator — Washington State University
Locations (1):
- Washington State University, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No
The investigators are not collaborating with other researchers, thus there is no plan to make IPD available.